CLINICAL TRIAL: NCT03000192
Title: HORIZONS: a Cohort Study to Explore Recovery of Health and Well-being in Adults Diagnosed With Cancer
Brief Title: HORIZONS: Understanding the Impact of Cancer Diagnosis and Treatment on Everyday Life
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: RHM CAN1199
Record Dates: First submitted 2016-12-13; First posted 2016-12-21 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer Female; Breast Neoplasm; Non-Hodgkin's B-cell Lymphoma; Non-Hodgkin's Lymphoma, Adult High Grade; NonHodgkin Lymphoma; Diffuse Large B Cell Lymphoma; Diffuse Large Cell Lymphoma, Adult; Ovarian Cancer; Ovarian Neoplasm; Endometrial Cancer; Endometrial Neoplasms; Cervical Cancer; Cervical Neoplasm; Primary Peritoneal Carcinoma; Fallopian Tube Cancer; Fallopian Tube Neoplasms; Vulvar Cancer; Vulvar Neoplasms
Keywords: Survivorship; Cancer; Recovery; Self-management; Cohort
MeSH Terms: conditions — Breast Neoplasms; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Fallopian Tube Neoplasms; Vulvar Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Breast cancer: Women aged <50 years
- Gynaecological cancers: Includes: cervical cancer, endometrial cancer, ovarian cancer, fallopian tube cancer, primary peritoneal cancer and vulval cancer
- Non-Hodgkin Lymphoma: Diffuse large B cell

SUMMARY:
The purpose of this study is to invite all people diagnosed with cancer who meet the eligibility criteria to complete questionnaires before their treatment begins and at regular intervals over time to assess the impact of cancer and its treatment on people's lives in the short, medium and long term. We will explore a range of factors to determine their role in both recovery of health and well-being and self-management. Although it is known that people who have had cancer are likely to experience a number of physical and psychological problems as a result of the disease and treatment, it is not known what the 'typical' course of recovery of health and well-being looks like, how long it takes and how this can be influenced. We will determine pathways to recovery of health and well-being following cancer diagnosis (initially breast cancer diagnosed <50 years, Non-Hodgkin Lymphoma and gynaecological cancers) and identify what factors influence this. This includes assessing the relative importance of the person's illness, personal attributes, perceived burden of treatment, role of the environment they live in, including health / social care and personal networks of support, and their ability and capacity to self-manage. We will identify who is most at risk of problems and what environmental supports and resources people are able to mobilise to support their self-management. We will also explore who has the confidence and ability to manage during and beyond treatment and what factors influence this and whether this leads to earlier problem resolution and restoration of health and well-being. This knowledge will be used to develop and test future supportive interventions to enhance the rapid recovery of health and well-being - our long term aim being to design ways of helping people with cancer in areas we identify as problematic for them.

ELIGIBILITY:
OVERALL ELIGIBILITY CRITERIA:

Inclusion Criteria:

* Have a new diagnosis of one of the selected cancer types determined through clinical assessment, cytology, histology or imaging or
* Have new / second primary cancer at a site previously treated for cancer
* Be awaiting primary curative intent treatment, including neoadjuvant treatment
* Be ≥16 years old.
* Be able to complete questionnaires in English
* Be able to provide written, informed consent

Exclusion Criteria:

* They do not have one of the specified cancer types
* Disease is recurrence / progression (either locally advanced or metastatic) at an existing cancer site
* They are having treatment for a potentially curative recurrence of disease e.g. locally advanced disease (i.e. they have been previously treated for the same cancer)
* They have metastatic disease from a cancer at another site (Previous diagnosis of cancer at any other site would not be grounds for exclusion unless disease was metastatic)
* They have synchronous primary cancers involving two or more of the HORIZONS specified cancer types (Please exclude synchronous gynaecological primary cancers, synchronous breast and gynaecological primary cancers, synchronous breast and non-Hodgkin's lymphoma primary cancers and synchronous non-Hodgkin's lymphoma and gynaecological cancers)

COHORT-SPECIFIC ELIGIBILITY CRITERIA:

BREAST CANCER COHORT

Inclusion:

* Women aged under 50 years old
* Stage 1, 2 or 3 breast cancer
* Have no distant metastases
* Patients due to undergo neoadjuvant treatment should be approached before this starts

For those whose core biopsy shows ductal carcinoma in situ (DCIS) only but post-excision biopsy pathology confirms invasive cancer, approach should be made as soon as possible following diagnosis and completion of the baseline questionnaire should be prior to the start of adjuvant treatment

Exclusion:

* Confirmed diagnosis of CIS (ductal or lobular) only
* Men

NON-HODGKIN LYMPHOMA COHORT

Inclusion:

* Any pathological diagnosis of Diffuse Large B Cell lymphoma (DLBCL) including;
* Secondary transforming or transformed DLBCL which has transformed from an indolent/low grade lymphoma (most commonly Follicular Lymphoma) as long as the low grade lymphoma was not treated and this is a recent transformation for which curative intent treatment has not yet started.
* Rare sub-types such as T cell rich Large B Cell Lymphoma and primary mediastinal (thymic) large B-cell lymphoma

Patients who have started steroid pre-phase treatment are eligible for approach before the start of chemotherapy.

GYNAECOLOGICAL CANCERS COHORT

ALL GYNAECOLOGICAL CANCERS

Gynaecological Cancer Exclusion criteria:

Synchronous gynaecological primary cancers. For example, synchronous ovarian and endometrial primary cancers.

OVARIAN CANCER SUB-COHORT

Ovarian Inclusion criteria:

Have a confirmed diagnosis either from cytology, histology, imaging or diagnostic primary surgery of either;

* Epithelial ovarian cancer including primary peritoneal cancer; fallopian tube cancer
* Ovarian carcinosarcoma
* Granulosa tumour of the ovary
* Patients should be entered prior to any treatment including surgery. However, where the diagnosis is only made at the time of surgery, these women may enter the study following surgery. Approach should be made as soon as possible following diagnosis and completion of the baseline questionnaire should occur prior to the start of adjuvant treatment.
* FIGO Stages: IA, IB, IC1, IC2, IC3, IIA, IIB, IIIA1

Ovarian Exclusion criteria:

* Borderline ovarian cancer
* Germ cell tumour
* Sarcoma

ENDOMETRIAL CANCER SUB-COHORT

Endometrial Inclusion criteria:

Have a confirmed diagnosis either from cytology, histology or imaging of;

* endometrial cancer
* endometrial carcinosarcoma

Patients should be entered prior to any treatment including surgery. However, where the diagnosis is only made at the time of surgery, these women may enter the study following surgery. Approach should be made as soon as possible following diagnosis and completion of the baseline questionnaire should occur prior to the start of adjuvant treatment.

- International Federation of Gynecology and Obstetrics (FIGO) Stages: IA, IB, II, IIIA, IIIB, IIIC1, IIIC2

Endometrial Exclusion criteria

* Choriocarcinoma
* Germ cell tumour
* Sarcoma

CERVICAL CANCER SUB-COHORT

Cervical Inclusion criteria:

Have a confirmed diagnosis either from cytology, histology or imaging of;

- Cervical cancer FIGO Stages: IA2, IB1, IB2, IIA1, IIA2, IIB, IIIA, IIIB

Cervical Exclusion criteria:

* FIGO stage IA1
* Cervical carcinoma in situ (CIS)
* Sarcoma
* Small cell cancer of the cervix

VULVAL CANCER SUB-COHORT

Vulval Inclusion criteria:

Have a confirmed diagnosis either from clinical assessment, cytology, histology, imaging of;

* Vulval cancer
* FIGO stages IA, IB, II, IIIA, IIIB, IIIC

Vulval Exclusion criteria:

* Basal cell carcinoma
* Melanoma
* Sarcoma
* Vulval intra-epithelial neoplasia (VIN)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The aim is to recruit people diagnosed with non-metastatic cancer through their clinical teams prior to primary treatment. Participants will be identified and recruited from NHS treatment centres across the UK, with centres chosen from those who express an interest through the Cancer Research Network (CRN) or directly to the HORIZONS Coordinating Centre. Centres will be selected for their proven research capability in these cancer types. Centres will indicate that they can approach a total sample of eligible patients and before treatment begins. Additionally, Centres will be selected to ensure the Study covers a wide range of geographical locations across England, Scotland, Wales and Northern Ireland, ethnically diverse populations and varying-sized hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Quality of Life in Adult Cancer Survivors (QLACS) | Change from Baseline (pre-treatment) up to 5 years [Anticipated]
  Primary outcome measure which assesses the quality of life in adult cancer survivors. It is comprised of 12 domains regarding cancer survivorship: generic (pain, fatigue, positive and negative feelings, cognitive and sexual problems, social avoidance) and cancer-specific (financial problems, family distress, recurrence distress, appearance concerns, benefits from cancer).
  Changes will be assessed at the following time-points:
  * Baseline (following diagnosis but pre-treatment)
  * 3 months after baseline (to monitor early adaptation and coping)
  * 12 months after baseline (to monitor coping and further adaptation)
  * 18 months after baseline (to explore early stages of recovery)
  * 24 months after baseline and further annual assessments (to monitor consequences in the longer term and how they are managed)

SECONDARY OUTCOMES:
EuroQoL 5 Dimensions 5 Levels (EQ-5D-5L) & Visual Analogue Scale (VAS) | Change from Baseline (pre-treatment) up to 5 years [Anticipated]
  Assesses health status for clinical and economic appraisal. Includes five domains: mobility, self-care, usual activities, pain/discomfort, anxiety/depression and five levels of severity.
EORTC-QLQ-C30 | Change from Baseline (pre-treatment) up to 5 years [Anticipated]
  Captures the impact of cancer and its treatment with 30 items assessing function (physical, role, cognitive, emotional, and social), symptoms (e.g. fatigue, pain, and nausea and vomiting) as well as global health and QoL.
EORTC Site Specific Modules: EORTC-QLQ -BR23, -CX24, -EN24, -NHL-HG29, -OV28, VU34 | Change from Baseline (pre-treatment) up to 5 years [Anticipated]
  Site-specific modules included to capture disease-specific consequences for Breast, Cervical, Endometrial, Ovarian and Vulval cancers, as well as High Grade Non-Hodgkin's Lymphoma (NHL). Modules will be supplemented with additional items from the EORTC item library to assess consequences not otherwise captured.
Hospital Anxiety and Depression Scale (HADS) | Change from Baseline (pre-treatment) up to 5 years [Anticipated]
  Comprises of 14 items with two 7-item subscales assessing anxiety and depression symptoms.
Medical Outcomes Study Social Support Survey (MOS-SSS) | Change from Baseline (pre-treatment) up to 5 years [Anticipated]
  Assesses the level of social support available and covers 4 domains (emotional/informational, tangible, affectionate support and positive social interaction).
Self-efficacy for Managing Chronic Disease (SEMCD) scale & Cancer Survivors' Self-Efficacy Scale (CS-SES) | Change from Baseline (pre-treatment) up to 5 years [Anticipated]
  SEMCD evaluates self-efficacy among patients with chronic medical conditions; whilst the CS-SES examines self-efficacy with reference to cancer-specific issues.

CONTACTS AND LOCATIONS:
Locations (111):
- United Kingdom (111):
  - Bronglais General Hospital, Aberystwyth
  - Monklands Hospital, Airdrie
  - Antrim Hospital, Antrim
  - William Harvey Hospital, Ashford
  - Wansbeck General Hospital, Ashington
  - Tameside Hospital, Ashton
  - University Hospital Ayr, Ayr
  - Ysbyty Gwynedd, Bangor
  - Basildon Hospital, Basildon
  - Basingstoke and North Hampshire Hospital, Basingstoke
  - Royal United Hospital, Bath
  - Bedford Hospital, Bedford
  - Arrowe Park Hospital, Birkenhead
  - Clatterbridge Hospital, Birkenhead
  - Birmingham City Hospital, Birmingham
  - Royal Blackburn Hospital, Blackburn
  - Pilgrim Hospital, Boston
  - Bradford Hospital, Bradford
  - Royal Sussex County Hospital, Brighton
  - Bristol Royal Infirmary, University Hospital Bristol, Bristol
  - Burnley General Teaching Hospital, Burnley
  - Kent and Canterbury Hospital, Canterbury
  - University Hospital of Wales, Cardiff
  - North Cumbria University Hospital, Carlisle
  - Epsom & St Helier Hospital, Carshalton
  - The Royal Marsden Hospital, Chelsea
  - Colchester General Hospital, Colchester
  - Queen Alexandra Hospital, Cosham
  - Northumbria Specialist Emergency Care Hospital, Cramlington
  - Leighton Hospital, Crewe
  - North Manchester General Hospital, Crumpsall
  - Darent Valley Hospital, Dartford
  - Royal Derby Hospital, Derby
  - Russells Hall Hospital, Dudley
  - Dumfries and Galloway Royal Infirmary, Dumfries
  - Ninewells Hospital, Dundee
  - Ulster Hospital, Dundonald
  - Hairmyres Hospital, East Kilbride
  - Eastbourne District General Hospital, Eastbourne
  - Western General Hospital, Edinburgh
  - Whipps Cross University Hospital, Epping
  - Queen Elizabeth Hospital, Gateshead
  - Medway Maritime Hospital, Gillingham
  - Beatson West Scotland Cancer Centre, Glasgow
  - James Paget University Hospital, Great Yarmouth
  - Royal Surrey County Hospital, Guildford
  - Calderdale Royal Hospital, Halifax
  - Charing Cross Hospital, Hammersmith
  - Hammersmith Hospital, Hammersmith
  - Northwick Park Hospital, Harrow
  - Conquest Hospital, Hastings
  - Withybush District General Hospital, Haverfordwest
  - Churchill Hospital, Headington
  - Hexham General Hospital, Hexham
  - Hillingdon Hospital, Hillingdon
  - Huddersfield Royal Infirmary, Huddersfield
  - Raigmore Hospital, Inverness
  - Ipswich Hospital, Ipswich
  - West Middlesex University Hospital, Isleworth
  - University Hospital Crosshouse, Kilmarnock
  - Queen Elizabeth Hospital, Kings Lynn
  - St James' Hospital, Leeds
  - Lincoln County Hospital, Lincoln
  - St John's Hospital, Livingston
  - University Hospital Llandough, Llandough
  - Royal Glamorgan Hospital, Llantrisant
  - St Bartholomew's Hospital, London
  - University College London Hospital, London
  - Macclesfield Hospital, Macclesfield
  - Maidstone Hospital, Maidstone
  - Manchester Royal Infirmary, Manchester
  - Saint Mary's Hospital, Manchester
  - The Christie Hospital, Manchester
  - Queen Elizabeth the Queen Mother Hospital, Margate
  - Borders General Hospital, Melrose
  - Newcastle Freeman Hospital, Newcastle
  - North Tyneside General Hospital, North Shields
  - Norwich University Hospital, Norwich
  - Nottingham University Hospitals NHS Trust - City Hospital Campus, Nottingham
  - Royal Oldham Hospital, Oldham
  - Peterborough City Hospital, Peterborough
  - Derriford Hospital, Plymouth
  - Royal Preston Hospital, Preston
  - East Surrey Hospital, Redhill
  - Ysbyty Glan Clwyd Hospital, Rhyl
  - Salford Royal, Salford
  - Salisbury District Hospital, Salisbury
  - Scarborough Hospital, Scarborough
  - Royal Hallamshire Hospital, Sheffield
  - Wexham Park Hospital, Slough
  - Ealing Hospital, Southall
  - Southampton General Hospital, University Hospital Southampton, Southampton
  - Southend University Hospital, Southend
  - St Albans City Hospital, St Albans
  - Royal Stoke University Hospital, Stoke-on-Trent
  - St Helier Hospital, Sutton
  - The Royal Marsden Hospital (Surrey), Sutton
  - King's Mill Hospital, Sutton in Ashfield
  - Musgrove Park Hospital, Taunton
  - St George's Hospital, Tooting
  - Royal Cornwall Hospital, Truro
  - Watford General Hospital, Watford
  - New Cross Hospital, Wednesfield
  - Sandwell General Hospital, West Bromwich
  - Weston General Hospital, Weston-super-Mare
  - West Cumberland Hospital, Whitehaven
  - Royal Hampshire County Hospital, Winchester
  - University Hospital Wishaw, Wishaw
  - Wrexham Maelor Hospital, Wrexham
  - Wythenshawe Hospital, Wythenshawe
  - York Teaching Hospital, York

IPD SHARING:
Plan to Share IPD: Yes
We encourage and facilitate data sharing by researchers from all disciplines.
  More detail can be found on our website: http://horizons-hub.org.uk/access_data.html
  If you have further questions about this process please contact us on 023 8059 6885 or msrg@soton.ac.uk.

REFERENCES:
- [Derived] Foster C, Calman L, Richardson A, May CR, Rogers A, Smith PW. HORIZONS protocol: a UK prospective cohort study to explore recovery of health and well-being in adults diagnosed with cancer. BMJ Open. 2019 Jul 26;9(7):e029662. doi: 10.1136/bmjopen-2019-029662. PMID 31350251